CLINICAL TRIAL: NCT05070481
Title: Clinical Observational and Statistical Study for Detection of Prevalence and Risk Factors of Disruptive Behavior in Children With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Prevalence of Disruptive Behavior in Children With Attention Deficit Hyperactivity Disorder(ADHD)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Eman Sayed Hassan Mahros (Other)
Responsible Party: Sponsor-Investigator, Eman Sayed Hassan Mahros, Principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 271087
Record Dates: First submitted 2021-09-18; First posted 2021-10-07 (Actual); Last update posted 2021-10-07 (Actual); Status verified 2021-09

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Identification of prevalence and Risk factors for disruptive behavior in children with Attention Deficit Hyperactivity Disorder and Early recognition of disruptive behavior in children with ADHD

DETAILED DESCRIPTION:
ADHD is asustaible pattern of inattention Hyperactivity and lmpulsive behavior which can have harmful consequences for the patients social life it was called childhood hyperkinetic reaction before it is estimated that 3 to 5 percent of children show symptoms in primary school in addition to the role of genetic factor in the incidence of this mental disorder ,family imbalance and other anxiety factors play arole in the continuity of disorder.disruptive behavior with a prevalence of 1 to 10percent is a prevalent disorder in primary school similar to ADHD it is 4 to 12 times more frequent among boys compared with girls . disruptive behavior characterized by aggression and violating others rights . This study is screening survey questionnaire study will be done in Assuit University children hospital Neuro psychiatric outpatient clinic in all children under 18 years old have ADHD and exclude other psychiatric problems as :Autism , depression , Schizophrenia or mental retardation . investigator will take full history : personal history : name , date of birth ,age,sex ,age of onset of ADHD ,type of ADHD,severity of ADHD ,type of disruptive behavior , history of treatment,Family history : sibling have ADHD,smoking of parents,drug use parents,social problems: divorce or death of parents . Investigator will use DSM V criteria as adignostic criteria and screening data evaluated by ADHD symptoms check list -4 (ADHD -sc4 scale scores) : symptoms count scores and symptoms severity scores . All for detect outcome of the patient with ADHD .

ELIGIBILITY:
Inclusion Criteria:

* All children under 18 years old with ADHD at Neuro pyshictric outpatient clinic

Exclusion Criteria:

* Any psychiatric problems other than ADHD like :Autism, depression, schizophrenia or mental retardation

Ages: 6 Months to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patient with ADHD that meet the selection criteria in the period from October 2021 till June 2022
Sampling Method: Probability Sample
Enrollment: 3 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of prevalence of disruptive behavior in children with ADHD by Sc -4 scale and DSM V score | Primarily from October 2021 till June 2022
  Screening data by ADHD symptoms chick list -4 rating scale(ADHD Sc-4 scale ) to detect symptoms count score and also invistigator use Diagnostic and Statistical Manual of mental disorders fifth edition(DSM V score) to assess the severity of symptoms

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Austerman J. ADHD and behavioral disorders: Assessment, management, and an update from DSM-5. Cleve Clin J Med. 2015 Nov;82(11 Suppl 1):S2-7. doi: 10.3949/ccjm.82.s1.01. PMID 26555810